CLINICAL TRIAL: NCT01797809
Title: Qlaira® Regulatory Post Marketing Surveillance Study in Korea
Brief Title: Qlaira rPMS (Regulatory Post Marketing Surveillance) Study in Korea
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16344; QL1212KR (Other: Company internal)
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-03

CONDITIONS: Contraception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: EV/DNG (Qlaira, BAY86-5027)

INTERVENTIONS:
Drug: EV/DNG (Qlaira, BAY86-5027) — Patients in daily life clinical practice tratment receiving Qlaira according to indication on the label.

SUMMARY:
The objective of this PMS is to gain information about safety and efficacy in real practice as a regulatory commitment required by KFDA (Korea Food and drug administration)

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Women after menarche and before menopause
* Women requesting contraception or Women diagnosed by a physician as having HMB due to non-organic cause who are also requesting contraception
* Women who are prescribed Qlaira® for the first time, during the study period

Exclusion Criteria:

- All contraindications according to the local marketing authorization have to be considered.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Generally healthy women after menarche and before menopause desiring contraception with or without HMB will be recruited who are determined to start Qlaira
Sampling Method: Non-Probability Sample
Enrollment: 757 (Actual)
Dates: Start 2013-05-11 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-05-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) including serious adverse events (SAEs) and Adverse Drug Reactions (ADRs) | Up to 6 months

SECONDARY OUTCOMES:
Contraceptive Efficacy by Number of unintended pregnancies | From 3 to 6 months
Contraceptive Efficacy by Compliance with Qlaira taking : Administered tablet number/prescribed tablet number | From 3 to 6 months
The relief of heavy menstrual bleeding symptom also will be calculated as an efficacy variable from admission to the study until final visit by subject's assessment | From 3 to 6 months
Number of subjects with improved heavy menstrual bleeding | From 3 to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, South Korea